CLINICAL TRIAL: NCT06496282
Title: The Efficacy of Lemborexant Versus Placebo on Improving Sleep Quality Among Hospital Rotating Shift Workers: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Lemborexant on Improving Sleep Quality Among Hospital Rotating Shift Workers
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Silpakorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEMY-2024
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Sleep
Keywords: Shift workers; Improving sleep; Lemborexant; Orexin receptor antagonists; Hospital rotating shift workers; Rotating shift workers
MeSH Terms: interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lemborexant 5 mg (Experimental): Lemborexant 5 mg 1 tab hs before bedtime
  Interventions: Drug: Lemborexant
- Placebo (Placebo Comparator): Placebo of Lemborexant 5 mg 1 tab hs before bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant — The participants will receive lemborexant for improving sleep quality at lease 30 days in 6 weeks of study
  Other Names: Dayvigo
  Arms: Lemborexant 5 mg
Drug: Placebo — The participants will receive placebo for improving sleep quality at lease 30 days in 6 weeks of study
  Other Names: Dayvigo placebo
  Arms: Placebo

SUMMARY:
Shift Work Sleep Disorder (SWSD) are caused by working shifts with a wake-up schedule and sleeping in a way that is different from the natural way of sleeping and avoiding sleep usually results in deviations. of the biological clock (Biological clock), which is an important cause of sleep problems including insomnia, excessive sleepiness or daytime sleepiness these problems was associated cadiovascular events, decrease quality of life and long term working. At the present there are limited information regarding the effectiveness of medications used to promote sleep in shift workers. Lemborexant is specific in binding to orexin type 2, which has a direct effect on sleep. and there are limited biomarkers monitoring from the use of lemborexant including still not found. Which studies have followed depressive symptoms, anxiety symptoms and cognition from a group of people with insomnia, the aim of study to assessment effectiveness of lemborexant on sleep efficiency, quality of life, symptoms of depression, cognition, BDNF, CRP, IL-6 and TNF-alpha levels. of volunteers working on rotating shifts.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* Rotating shift workers at least 3 months and continue rotating shift until end of study
* Participants who have sleep problem especially total sleep time lower than 6 hours and/or unable to sleep effectively according to the ICSD-3 at least 1 criteria
* Participants who have sleepy while working and have Epworth sleepiness scale in shift grater than or equal to 10 points

Exclusion Criteria:

* Receiving drug interaction esp. drugs induced CYP3A4 (moderate to severe) or drugs inhibited CYP3A4 (moderate to severe)
* Untreatment mental health disease or in process medication adjustment
* Hepatic function in Chid-Pugh C
* Pregnancy
* Breastfeeding
* Participants who in process medication adjustment such as mental heat, neurology, insomnia, contraceptive drugs.
* Diagnosis obstructive sleep apnea (OSA) with or without CPAP using or diagnosis restless leg syndrome or circadian rhythm disorders or narcolepsy
* Complex sleep behaviors such as sleep driving, sleep phone, sleep cooking
* HAM-D grater than or equal to 24 points
* HAM-A grater than or equal to 24 points
* Caffeine taking grater than 400 mg/day or can't not hold caffeine 4 hours before bedtime
* Substance abuse or alcoholism within 2 years ago
* Alcohol intake grater than 140 g of alcohol per week in female or intake grater than 210 g of alcohol per week in male or can't control alcohol drinking greater than 20 g of alcohol per day or can't hold alcohol within 3 hours before bedtime
* Cannabinoid using within 1 week ago
* Participants who have underlying disease such as stroke, atrial fibrillation, chronic obstructive pulmonary disease, hepatic impairment, severe renal impairment, cognitive impairment, cancer, chronic pain
* Participant who use of benzodiazepine or non-benzodiazepine in treatment of insomnia
* Participant who have nocturia problem
* Participant who have mental health problem which the physician conclude it affect the safety of participant
* Participant who have suicidal thinking with or without plan or have suicidal behaviors within 10 years ago
* Participant who have major surgery schedule during the study
* Travel across greater than 3 time zone within 2 weeks before include participant
* Allergy of lemborexant or component of lemborexant
* Have previously participated in study that used lemborexant
* Participant who

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Assessment effective of sleep quality in lemborexant 5 mg compare with placebo group | 1 week after screening, 3 and 6 weeks after lemborexant administration
  Sleep quality improvement evaluated by physician with actigraphy (Fitbit inspire 2) after lemborexant administration in 3 and 6 week.
Changing of Brian-derived neurotropic (BDNF) in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Blood sample of BDNF changing in 1 week after screening and 6 weeks after lemborexant administration

SECONDARY OUTCOMES:
Assessment effective of sleepiness level in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Sleepiness level improvement evaluated by physician with Epworth sleepiness scale after lemborexant administration in 1 week after screening and 6 weeks after lemborexant administration
Assessment effective of sleep quality in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Sleep quality improvement evaluated by physician with Pittsburgh sleep quality index (PSQI) in 1 week after screening and 6 weeks after lemborexant administration
Assessment of depression symptoms in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Depression symptoms improvement evaluated by physician with Hamilton depression rating scale (HAM-D) after lemborexant administration in 1 week after screening and 6 weeks after lemborexant administration
Assessment of anxiety symptoms in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Anxiety symptoms improvement evaluated by physician with Hamilton anxiety rating scale (HAM-A) after lemborexant administration in 1 week after screening and 6 weeks after lemborexant administration
Assessment of cognition in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Cognition improvement evaluated by physician with Motreal cognitive assessment (MOCA), Grooved pegboard test and Digit symbol substitution test in1 week after screening and 6 weeks after lemborexant administration
Assessment of quality of life in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Quality of life improvement evaluated by physician with EuroQOL five dimensions questionnaires (EQ-5D )in 1 week after screening and 6 weeks after lemborexant administration
Changing of CRP, IL-6 and TNF-alpha in lemborexant 5 mg compare with placebo group | 1 week after screening and 6 weeks after lemborexant administration
  Blood sample of CRP, IL-6 and TNF-alpha changing in 1 week after screening and 6 weeks after lemborexant administration

CONTACTS AND LOCATIONS:
Overall Officials: Tipvilai Taweepunturat, Pharm.D., Study Chair — Faculty of Pharmacy Siam University; Abisith Dechachongjumroen, MD, Principal Investigator — Phramongkutklao hospital and College of Medicine; Wananwat Danworapong, MD, Principal Investigator — Phramongkutklao hospital and College of Medicine; Juthathip Suphanklang, BCP, Study Director — Phramongkutklao hospital and College of Medicine; Pasiri Sithinamsuwan, MD, Study Director — Phramongkutklao hospital and College of Medicine
Locations (1):
- Phramongkutklao Hospital, Ratchathewi, Bangkok, Thailand